CLINICAL TRIAL: NCT02170688
Title: Use of Electrical Impedence to Measure Lean Body Weight as a Determinant of the Dose of Contrast Media for Abdominal CT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pro00010850
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: IV Contrast Dosing
Keywords: IV contrast; contrast dosing
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- Fixed dose (Active Comparator): 50 subjects will receive contrast media based on a fixed dose. Each will receive 125 mL of Isovue 370 (370 mg of iodine/mL) administered at 4 mL/sec (1.48 gmI/sec for 31.25 sec).
  Interventions: Drug: Isovue 370
- Total body weight (Active Comparator): 25 subjects will receive contrast media dose based on the total body weight. Total body weight will be determined. Both men and women will receive contrast media at a dose of 0.7 gmI/kg (1.78 mL of Isovue 370/kg) or 0.30 gmI/lb (0.81 mL of Isovue 370/lb). The injection rate will be 0.058 mL/sec/kg (0.026 mL/sec/lb).
  Interventions: Drug: Isovue 370; Other: Weight calculation
- Calculated lean body weight (Active Comparator): 25 subjects will receive contrast media dose based on the calculated lean body weight. Total body weight and height will be determined. From this data the lean body weight will be calculated.
  Men will receive a dose of 0.86 gmI / kg LBW (2.32 mL of Isovue 370/kg at 0.074 mL/sec/kg) or 0.39 gmI/lb LBW (1.05 mL of Isovue 370/lb at 0.034 mL/sec/lb). Women will receive a dose of 0.92 gmI/kg LBW (2.49 mL of Isovue 370/kg at 0.080 mL/sec/kg) or 0.42 gmI/lb LBW (1.13 mL of Isovue 370/kg at 0.036 mL/sec/kg).
  Interventions: Drug: Isovue 370; Other: Weight calculation
- Measured lean body weight (Active Comparator): 50 subjects will receive contrast media dose based on the measured lean body weight. Lean body weight will be determined using the Tanita body composition/analyzer scales. From this data the lean body weight will be calculated.
  Men will receive a dose of 0.86 gmI / kg LBW (2.32 mL of Isovue 370/kg at 0.074 mL/sec/kg) or 0.39 gmI/lb LBW (1.05 mL of Isovue 370/lb at 0.034 mL/sec/lb). Women will receive a dose of 0.92 gmI/kg LBW (2.49 mL of Isovue 370/kg at 0.080 mL/sec/kg) or 0.42 gmI/lb LBW (1.13 mL of Isovue 370/kg at 0.036 mL/sec/kg).
  Interventions: Drug: Isovue 370; Other: Weight calculation
- Estimated lean body (eLBW) weight (Active Comparator): 25 subjects will receive contrast media dose based on the estimated lean body (eLBW) weight. Estimated lean body weight will be determined by using a unique software program which measures the sum of the posterior to anterior attenuation from the digital scout radiograph (abbreviated as sqrt PA) obtained during the standard planning scan of the abdominal/pelvic CT. Men will receive a dose of 0.86 gmI / kg eLBW (2.32 mL of Isovue 370/kg at 0.074 mL/sec/kg) or 0.39 gmI/lb eLBW (1.05 mL of Isovue 370/lb at 0.034 mL/sec/lb). Women will receive a dose of 0.92 gmI/kg eLBW (2.49 mL of Isovue 370/kg at 0.080 mL/sec/kg) or 0.42 gmI/lb eLBW (1.13 mL of Isovue 370/kg at 0.036 mL/sec/kg).
  Interventions: Drug: Isovue 370; Other: Weight calculation

INTERVENTIONS:
Drug: Isovue 370 — All contrast media doses administered for this study are within the FDA approved dose range in the package insert.
Other: Weight calculation
  Arms: Calculated lean body weight; Estimated lean body (eLBW) weight; Measured lean body weight; Total body weight

SUMMARY:
There are several different methods that can be used to determine the dose of iodinated contrast material for a CT scan. These include a standard fixed dose, a dose based on total body weight, a dose based on body mass index, a dose based on lean body weight, and a dose based on estimated lean body weight. The fixed dose method uses a predetermined amount of contrast material for all patients having a CT scan of the abdomen regardless of size. This is the standard procedure currently used at Duke. The other methods use the patient's weight, either the total body weight or lean body weight, to determine the amount of contrast necessary for the CT exam. For this study, the investigators will use the fixed dose, total body weight, the lean body weight, and estimated lean body weight methods. The purpose of this study is to evaluate these five methods of determining the IV contrast volume and which may be best for abdominal CT scanning.

ELIGIBILITY:
Inclusion Criteria:

* male or non-lactating, non-pregnant females
* 18 years or older who are able to give written informed consent

Exclusion Criteria:

* a chronic underlying liver disease such as cirrhosis, fatty infiltration of the liver or glycogen storage diseases
* patients with a prolonged cardiac transit time such as those with a congested heart failure, a history of prior cardiac valve replacement, or restrictive/constrictive pericarditis
* patients having undergone any other radiological procedure utilizing iodinated contrast with the 24 hours prior to the CT exam
* patients above a certain total body weight (440 lbs.) due to limitation of the scales themselves (determined by manufacturer)
* any subjects with a history of hypersensitivity to iodine-containing compounds or renal insufficiency (serum creatinine >1.8)
* subjects with implanted electronic devices (pacemakers, defibrillators, insulin pumps, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2004-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ho, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Body Weight: 25 subjects will receive contrast media dose based on the total body weight. Total body weight will be determined. Both men and women will receive contrast media at a dose of 0.7 gmI/kg (1.78 mL of Isovue 370/kg) or 0.30 gmI/lb (0.81 mL of Isovue 370/lb). The injection rate will be 0.058 mL/sec/kg (0.026 mL/sec/lb).
  Isovue 370: All contrast media doses administered for this study are within the FDA approved dose range in the package insert.
  Weight calculation
- Calculated Lean Body Weight: 25 subjects will receive contrast media dose based on the calculated lean body weight. Total body weight and height will be determined. From this data the lean body weight will be calculated.
  Men will receive a dose of 0.86 gmI / kg LBW (2.32 mL of Isovue 370/kg at 0.074 mL/sec/kg) or 0.39 gmI/lb LBW (1.05 mL of Isovue 370/lb at 0.034 mL/sec/lb). Women will receive a dose of 0.92 gmI/kg LBW (2.49 mL of Isovue 370/kg at 0.080 mL/sec/kg) or 0.42 gmI/lb LBW (1.13 mL of Isovue 370/kg at 0.036 mL/sec/kg).
  Isovue 370: All contrast media doses administered for this study are within the FDA approved dose range in the package insert.
  Weight calculation
- Measured Lean Body Weight: 50 subjects will receive contrast media dose based on the measured lean body weight. Lean body weight will be determined using the Tanita body composition/analyzer scales. From this data the lean body weight will be calculated.
  Men will receive a dose of 0.86 gmI / kg LBW (2.32 mL of Isovue 370/kg at 0.074 mL/sec/kg) or 0.39 gmI/lb LBW (1.05 mL of Isovue 370/lb at 0.034 mL/sec/lb). Women will receive a dose of 0.92 gmI/kg LBW (2.49 mL of Isovue 370/kg at 0.080 mL/sec/kg) or 0.42 gmI/lb LBW (1.13 mL of Isovue 370/kg at 0.036 mL/sec/kg).
  Isovue 370: All contrast media doses administered for this study are within the FDA approved dose range in the package insert.
  Weight calculation
- Estimated Lean Body (eLBW) Weight: 25 subjects will receive contrast media dose based on the estimated lean body (eLBW) weight. Estimated lean body weight will be determined by using a unique software program which measures the sum of the posterior to anterior attenuation from the digital scout radiograph (abbreviated as sqrt PA) obtained during the standard planning scan of the abdominal/pelvic CT. Men will receive a dose of 0.86 gmI / kg eLBW (2.32 mL of Isovue 370/kg at 0.074 mL/sec/kg) or 0.39 gmI/lb eLBW (1.05 mL of Isovue 370/lb at 0.034 mL/sec/lb). Women will receive a dose of 0.92 gmI/kg eLBW (2.49 mL of Isovue 370/kg at 0.080 mL/sec/kg) or 0.42 gmI/lb eLBW (1.13 mL of Isovue 370/kg at 0.036 mL/sec/kg).
  Isovue 370: All contrast media doses administered for this study are within the FDA approved dose range in the package insert.
  Weight calculation
Period: Overall Study
Arm/Group | Fixed Dose | Total Body Weight | Calculated Lean Body Weight | Measured Lean Body Weight | Estimated Lean Body (eLBW) Weight
Started | 29 | 29 | 29 | 27 | 25
Completed | 25 | 26 | 25 | 25 | 25
Not Completed | 4 | 3 | 4 | 2 | 0
Not completed — Exclusion Criteria: Fatty Liver | 4 | 2 | 3 | 2 | 0
Not completed — Full dose not received | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose | Total Body Weight | Calculated Lean Body Weight | Measured Lean Body Weight | Estimated Lean Body (eLBW) Weight | Total
Number analyzed (Participants) | 29 | 29 | 29 | 27 | 25 | 139
Age, Customized [Number; unit: participants]
  ≥18 years | 29 | 29 | 29 | 27 | 25 | 139
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 10 | 13 | 12 | 61
  Male | 20 | 12 | 19 | 14 | 13 | 78
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 29 | 27 | 25 | 139

OUTCOME MEASURES:

1. Secondary Outcome: Difference in Volume of Contrast Used, Measured in Milliliters
Time Frame: baseline, post-dose imaging (approximately 1hr)
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Fixed Dose | Total Body Weight | Calculated Lean Body Weight | Measured Lean Body Weight | Estimated Lean Body (eLBW) Weight
Number analyzed (Participants) | 25 | 26 | 25 | 25 | 25
Milliliters | 125 (0) | 130 (32) | 139 (25) | 135 (28) | 105 (18)

2. Primary Outcome: Difference in Enhancement of the Liver and Blood Vessels Over Time, Measured in Hounsfield Units (HU)
Description: Operator-defined regions-of-interest (ROI) will be obtained from liver parenchyma, the portal vein and the abdominal aorta prior to contrast administration and on each slice through the liver post-contrast. Sum of all three areas reported as Summed measurement.
Time Frame: baseline, post-dose imaging (approximately 1hr)
Measure: Mean (Standard Deviation); unit: Hounsfield units (HU)
Arm/Group | Fixed Dose | Total Body Weight | Calculated Lean Body Weight | Measured Lean Body Weight | Estimated Lean Body (eLBW) Weight
Number analyzed (Participants) | 25 | 26 | 25 | 25 | 25
Hounsfield units (HU)
  Liver | 116 (15) | 124 (13) | 121 (14) | 120 (11) | 124 (12.6)
  Portal Vein | 158 (21) | 167 (24) | 164 (24) | 161 (17) | 183 (30.9)
  Aorta | 145 (18) | 152 (17) | 148 (18) | 145 (13) | 153 (20)
  Summed Measurement | 419 (50) | 443 (51) | 433 (50) | 426 (33) | 461 (56)

ADVERSE EVENTS:
Arm/Group | Fixed Dose | Total Body Weight | Calculated Lean Body Weight | Measured Lean Body Weight | Estimated Lean Body (eLBW) Weight
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes